CLINICAL TRIAL: NCT05101915
Title: Phase II Open Label Study of a Nebulised Nitric Oxide Generating Solution in Patients With Mycobacterium Abscessus Pulmonary Disease
Brief Title: Study of a Nebulised Nitric Oxide Generating Solution in Patients With Mycobacterium Abscessus
Acronym: NOMAB
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: TSC recommended early termination due to lack of futility of the trial.
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02702
Record Dates: First submitted 2021-09-13; First posted 2021-11-01 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis
Keywords: Mycobacterium abscessus
MeSH Terms: conditions — Cystic Fibrosis; Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Intervention Model Description: This is a single centre, non-randomized, open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Single arm trial involving all patients receiving IMP
  Interventions: Drug: RESP301

INTERVENTIONS:
Drug: RESP301 — Inhaled IMP delivered via nebulisation

SUMMARY:
* To evaluate the change in M. abscessus cfu/g in induced sputum samples from baseline to the end of treatment with RESP301 in patients with cystic fibrosis who have treatment-naïve or treatment-refractory M. abscessus-pulmonary disease
* To assess the safety and tolerability of RESP301 during treatment (28 days) and follow up (84 days) in patients with cystic fibrosis who have treatment naïve or treatment refractory M. abscessus-pulmonary disease

DETAILED DESCRIPTION:
Investigators will undertake an eighteen-week single centre, open label study in participants with cystic fibrosis infected with Mycobacterium abscessus (M. abscessus)-pulmonary disease (-PD).

The study will treat particpants with cystic fibrosis (CF) attending the Adult Cystic Fibrosis Centre at the Royal Papworth Hospital, Cambridge, United Kingdom. Participants will be consented and screened for the RESP301-003 study to enable approximately 12 participants to commence treatment with RESP301.

Participants will have M abscessus-PD as defined by the ATS/IDSA, specifically: (i) two or more positive sputum cultures for M. abscessus; (ii) radiological change consistent with NTM-PD; and (iii) symptoms consistent with NTM-PD, after exclusion of other causes.

Participants will be recruited who (1) have not commenced antibiotic treatment for M. abscessus-PD or (2) have treatment refractory M. abscessus-PD (defined as remaining sputum culture positive after 6 months or more of treatment). Treatment-refractory participants will be suitable for enrolment in the study if date of first dosing is at least 2 months since a change in M. abscessus treatment (or 4 months since change of Clofazimine).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of ≥18 years at time of informed consent
2. Patients with a clinical diagnosis of CF and confirmed by genetic testing
3. Diagnosis of treatment naïve or treatment refractory M. abscessus-PD
4. Signed informed consent documentation (indicating an understanding of the purpose and a willingness to meet the requirements for participation in the study)

Exclusion Criteria:

1. FEV1 <40% predicted
2. Methaemoglobin concentration > 2%
3. Use of nitric oxide donor medications such as prilocaine, sodium nitroprusside, and nitroglycerine within 30 days of proposed first treatment
4. Use of phosphodiesterase inhibitors (e.g., sildenafil) within 30 days of proposed first treatment
5. Evidence of pulmonary hypertension
6. History of frequent low volume or massive haemoptysis
7. Liver disease (i.e. liver cirrhosis, portal hypertension)
8. Subjects who have undergone organ transplantation
9. Pregnancy or lactation (female participants only)
10. Subjects who will not use appropriate forms of contraception for the duration of the study
11. Contraindication or unable to complete lung function testing
12. Contraindication or unable to tolerate nebulised hypertonic saline
13. Changes to previous NTM antibiotic regimen within two months of first dose of study treatment (or 4 months for clofazimine)
14. Subject has received investigational treatment as part of another interventional clinical trial within two months of the proposed first day of treatment
15. Required antibiotic treatment for a pulmonary exacerbation within 2 weeks of enrolment to the study.
16. Inability to undergo study related activities and / or commitments
17. Any subject who in the opinion of the investigator would not be best served by participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Mycobacterial load in induced sputum samples | Through study completion, average one year
  The primary efficacy endpoint is the change in mycobacterial load in induced sputum samples as assessed by log10 change in M. abscessus cfu/g sputum from Baseline to End of Treatment.
Safety and tolerability | Through study completion, average one year
  Safety and tolerability will be assessed by clinical safety laboratory measurements, physical examinations, vital signs, concomitant medications; cumulative incidence of adverse events (AEs), serious adverse events (SAEs) and severe AEs.

SECONDARY OUTCOMES:
Change in mycobacterial load in spontaneously expectorated daily sputum samples | Through study completion, average one year
  The change in mycobacterial load in spontaneously expectorated daily sputum samples from Baseline to Final Week of Treatment. For this secondary endpoint, Baseline is defined as the average M. abscessus cfu/g sputum in samples from the mornings of Days -14 to -1 inclusive. The final seven days of treatment are days 22 to 28 inclusive; the sputum samples are produced on the following mornings
Proportion of individuals achieving a ≥2 log10 decrease in the mycobacterial load - induced samples | Through study completion, average one year
  Proportion of individuals achieving a ≥2 log10 decrease in the mycobacterial load as assessed by change in M. abscessus cfu/g in the induced sputum samples from Baseline to End of Treatment.
Proportion of individuals achieving a ≥2 log10 decrease in the mycobacterial load - spontaneous samples | Through study completion, average one year
  Proportion of individuals achieving a ≥2 log10 decrease in the mycobacterial load as assessed by change in M. abscessus cfu/g in the spontaneously expectorated sputum samples from Baseline to Final Week of Treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom